CLINICAL TRIAL: NCT01178151
Title: Pilot Study of Everolimus in the Treatment of Neoplasms in Patients With Peutz-Jeghers Syndrome
Brief Title: Study of Everolimus in the Treatment of Advanced Malignancies in Patients With Peutz-Jeghers Syndrome
Acronym: EVAMP
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Heinz-Josef Klumpen, MD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMCmedonc010; 2010-020451-32 (EudraCT Number)
Record Dates: First submitted 2010-07-26; First posted 2010-08-10 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Peutz-Jeghers Syndrome; Neoplastic Processes; Neoplasm Metastasis
Keywords: Peutz-Jeghers syndrome; mTOR inhibition; cancer
MeSH Terms: conditions — Peutz-Jeghers Syndrome; Neoplastic Processes; Neoplasm Metastasis; Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- afinitor (Experimental): 10mg afinitor daily orally
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — 10mg daily orally
  Other Names: Afinitor, RAD001, everolimus

SUMMARY:
In this pilot study the investigators will treat all patients known with Peutz-Jeghers syndrome (PJS) who are diagnosed with advanced malignancies with everolimus 10mg daily until disease progression. Most patients with PJS have an inherited LKB1 mutation leading to aberrant m-TOR activity. Their risk to develop malignancies or intestinal polyps is probably related to this constitutive mTOR signaling. The hypothesis is that mTOR inhibition is an effective anticancer treatment in PJS patients with advanced malignancies.

ELIGIBILITY:
Tow cohorts of PJS patients will be included. Cohort 1: Advanced malignancy Cohort 2: High risk polyps

General inclusion criteria:

1. Known Peutz-Jeghers disease (with LKB1 mutation)
2. No concurrent systemic anti cancer treatment
3. No prior treatment with m-TOR inhibitor
4. Prior malignancies or concurrent second malignancies are allowed
5. Prior systemic therapy is permitted with a washout time of at least 4 weeks
6. ECOG/ WHO performance 0-2
7. Age > 18 years
8. Adequate renal function (defined as creatinine < 150 μmol/L)
9. Adequate liver function (bilirubin < 1.5 times upper limit of normal, ALAT or ASAT < 5.0 times upper limit of normal in case of liver metastases and < 2.5 the upper limit of normal in absence of liver metastases
10. Adequate bone marrow function (WBC > 3.0 x 10 9/L, platelets > 100 x 10 9/L)
11. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
12. No pregnancy or lactating and ifof childbearing potential patients must agree to use a reliable contraceptive method throughout the study
13. No serious concomitant systemic disorder that would compromise the safety of the patient,at the discretion of the investigator
14. Signed informed consent according to ICH/GCP.
15. No uncontrolled symptomatic hyperglycaemia

Specific inclusion criteria for cohort 1:

1. Cytological or histological confirmed carcinoma
2. Metastatic or non-resectable disease
3. Patients with clinically and/or radiographically documented measurable lesion according to

RECIST criteria:

1. X-ray, physical exam > 20 mm
2. Spiral CT scan > 10 mm
3. Non-spiral CT scan > 20 mm

Specific inclusion criteria for cohort 2:

1. Known high risk polyps (definition see page 19)
2. Ability to undergo endoscopies

Specific Exclusion criteria:

Symptomatic PJ-polyps, defined as polyps likely to be responsible/causal for the abdominal symptoms the patient presents with.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
To determine the response rate of Everolimus in patients with advanced cancer and PJS. | During treatment, expected avarage of 12 months
  Determined with regular radiological scans once every 9 weeks and measured following RECIST 1.1

SECONDARY OUTCOMES:
To determine the overall survival of PJS patients treated with everolimus for advanced malignancies | avarage of 18 months
  The time between date of entering the study and date of death will be collected.
To determine the time to progression of PJS patients treated with everolimus for advanced malignancies. | During treatment, expected avarage of 12 months
  Determined with regular radiological scans once every 9 weeks and measured following RECIST 1.1
To determine the safety and toxicity of Everolimus in this patient population | During treatment, expected avarage of 12 months
  Number of Participants with Adverse Events determined by the CTCAE 4.0 as a Measure of Safety and Tolerability
To determine if there is an association between measured drug blood levels and treatment outcome measured as response to treatment determined by RECIST | During treatment, expected avarage of 12 months
  Drug trough levels will be taken once every 3 weeks and stored frozen until measurement at the end of the study
To assess markers for activated mTOR pathway (including phospho-S6 and phospho-4E BP1) in all pre-treatment tissue specimens and collected specimens during treatment and correlate with response to treatment. | During treatment, expected avarage of 12 months
  All patients who are willing to undergo extra tissue collection will have a tumor and where possible a polyp biopsy before treatment and for tumor biopsy in week 2 and 4 and for polyps once every 6 months during treatment for biomarker investigations. The activity of mTOR and its downstream targets will be measured in the tumor as well as the arborization pattern and apoptosis activity in the polyps.

CONTACTS AND LOCATIONS:
Overall Officials: Heinz-Josef Klumpen, MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (2):
- Netherlands (2):
  - Academic Medical Center, Amsterdam
  - Erasmus Medical Center, Rotterdam

REFERENCES:
- [Derived] de Brabander J, Eskens FALM, Korsse SE, Dekker E, Dewint P, van Leerdam ME, van Eeden S, Klumpen HJ. Chemoprevention in Patients with Peutz-Jeghers Syndrome: Lessons Learned. Oncologist. 2018 Apr;23(4):399-e33. doi: 10.1634/theoncologist.2017-0682. Epub 2018 Jan 25. PMID 29371475